CLINICAL TRIAL: NCT02427048
Title: Adherence to Clinical Practice Guidelines and the Impact of Audit and Feedback in the Emergency Department
Brief Title: Clinical Practice Guidelines and Impact of Audit and Feedback in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15-0400
Record Dates: First submitted 2015-04-15; First posted 2015-04-27 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Shock, Septic; Community Acquired Pneumonia
Keywords: Clinical Practice Guidelines
MeSH Terms: conditions — Shock, Septic; Community-Acquired Pneumonia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-Intervention (No Intervention): Delayed feedback and peer comparison
- Feedback with Peer Comparison (Experimental): Individualized adherence feedback with peer comparison
  Interventions: Behavioral: Feedback with Peer Comparison

INTERVENTIONS:
Behavioral: Feedback with Peer Comparison — Email detailing adherence to CAP and SS CPG for every month since start of study. Physicians will be provided individualized feedback and given patient identifiers for each patient that received non-adherent care.
  Arms: Feedback with Peer Comparison

SUMMARY:
This study will develop and test an intervention given to emergency medicine providers to improve adherence to clinical practice guidelines (CPGs) for pneumonia and sepsis.

DETAILED DESCRIPTION:
This study will be performed at Denver Health Medical Center, a 477-bed urban, safety-net, acute-care hospital located in Denver, Colorado. The adult ED is staffed by board-certified emergency physicians at all times. These physicians supervise the care of all patients being managed by resident physicians, nurse practitioners, physician assistants, and medical students. Approximately 430 patients are admitted to the hospital from the ED each year with community-acquired pneumonia (CAP) and severe sepsis (SS).

Adherence to CPGs will be measured at the level of the attending emergency physician. All employed, attending emergency physicians working clinically in the adult ED at Denver Health Medical Center at the start of the study will be included.

The investigators will use a step-wedge design to randomize physicians into clusters. Randomization of physicians into clusters and randomization of clusters to intervention timing will occur one week prior to delivery of the intervention to cluster one. he intervention will consist of monthly audit and feedback on adherence to CPGs for CAP and SS. Once a cluster enters its first intervention month, all physicians in that cluster will receive an email detailing their adherence to both CAP and SS CPG for every month since the start of the study. Adherence to the entire CPG as well as each component of the CPG will be provided. In addition, physicians will be shown the median prevalence of adherence for all physicians as well as where their adherence ranks among their physician group. Lastly, in a separate secure email, physicians will be given patient identifiers (i.e., name, MRN, date of visit) for each patient that received non-adherent care and will be told which component of care was not adherent to the respective CPG so that they can review the case themselves, if desired.

ELIGIBILITY:
Inclusion Criteria:

* Attending emergency medicine physicians working clinically in the Adult Emergency Department at Denver Health Medical Center at the start of the study.

Exclusion Criteria:

* None. All eligible physicians will be included.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Adherence to Community-Acquired Pneumonia and Severe Sepsis Clinical Practice Guidelines | 30 days post-intervention and 60 days post-intervention
  Adherence will be determined via chart review of patients and will be measured by concordance with published clinical practice guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Trent, MD, Principal Investigator — Denver Health and Hospital Authority

IPD SHARING:
Plan to Share IPD: No